CLINICAL TRIAL: NCT03871478
Title: Comparing the Efficacy of Local Anesthetics in Mohs Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Richard J. MacKay Endowment Fund (Unknown); Benefactor Life Members' Research Grant (Unknown); The Ottawa Hospital Division of Dermatology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #20160131
Record Dates: First submitted 2019-03-01; First posted 2019-03-12 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Lidocaine; Bupivacaine; Mohs Surgery; Anesthetic
MeSH Terms: interventions — Lidocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lidocaine (Active Comparator): Buffered lidocaine 1% with epinephrine 1:200,000 Injected at the start of every Mohs excision stage
  Interventions: Drug: Lidocaine
- Bupivacaine (Active Comparator): Bupivacaine 0.5% with epinephrine 1:200,000 Injected at the start of every Mohs excision stage
  Interventions: Drug: Bupivacaine
- Lidocaine and Bupivacaine (Active Comparator): Buffered lidocaine 1% with epinephrine 1:200,000 and bupivacaine 0.5% with epinephrine 1:200,000 injected sequentially.
  Injected at the start of every Mohs excision stage
  Interventions: Drug: Lidocaine and Bupivacaine

INTERVENTIONS:
Drug: Lidocaine — See Arm Description
  Arms: Lidocaine
Drug: Bupivacaine — See Arm Description
  Arms: Bupivacaine
Drug: Lidocaine and Bupivacaine — See Arm Description
  Arms: Lidocaine and Bupivacaine

SUMMARY:
Mohs surgery is a very effective option in removing non-melanoma skin cancers, as the tissue being removed is analyzed the same day. If there are remnants of cancer cells in the tissue removed, the Mohs surgeon will go back and remove further tissue and repair the surgical wound all within the same day.

Unfortunately, postoperative pain is quite prevalent among patients requiring Mohs procedures, as up to 52% require an additional oral pain medication. Lidocaine is the most commonly used anesthetic used in Mohs given its rapid onset of action. However, the duration of lidocaine's effect is much shorter than bupivacaine, which may translate into increased postoperative pain.

To date, there are no specific studies comparing bupivacaine alone, lidocaine alone or both in conjunction in Mohs procedures.

The investigators predict bupivacaine alone and bupivacaine used in conjunction with lidocaine are more effective in managing pain during Mohs surgery than lidocaine alone.

To test our hypothesis, the investigators plan to have 105 patients receive either lidocaine alone, bupivacaine alone, or lidocaine and bupivacaine in conjunction during their Mohs procedure. Pain will be evaluated at various time points throughout the surgery.

DETAILED DESCRIPTION:
Mohs surgery is a very effective option in removing non-melanoma skin cancers, as the tissue being removed is analyzed the same day. If there are remnants of cancer cells in the tissue removed, the Mohs surgeon will go back and remove further tissue and repair the surgical One option for treating non-melanoma skin cancer is Mohs Surgery, also known as Mohs Micrographic Surgery or Mohs Procedure.

Mohs surgery is a full-day procedure where your skin cancer will be removed and processed immediately after in our lab. The investigators look at the edges of the skin that the investigators have removed to see if there is any cancer left. If any of the edges show that there is still cancer, the investigators go back and remove more. The investigators will repeat this process until all of the margins of your skin are clear from cancer. After all the cancer is removed, the investigators will reconstruct the area that has been removed to give you the best cosmetic and functional result.

Throughout this procedure, the investigators will inject local anesthetic or "freezing" to reduce the discomfort associated with skin cancer surgery. There are two different types of local anesthetic that the investigators are studying to reduce this pain. One anesthetic is called lidocaine and the other is bupivacaine. A third option is to use a combination of lidocaine and bupivacaine. Lidocaine and bupivacaine are both approved by Health Canada for its use in providing local anesthesia.

WHY IS THIS STUDY BEING DONE? The purpose of this study is to look at which of the approved interventions (lidocaine, bupivacaine or a combination of the two injected sequentially) works best to reduce pain during and after Mohs surgery.

HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY? It is anticipated that about 105 people will take part in this study from The Mohs Clinic at the Parkdale Dermatology Clinic of The Ottawa Hospital.

This study should take three months to complete and the results should be known in about 6 months.

ASSIGNMENT TO A GROUP If you decide to participate then you will be "randomized" into one of the groups described below. Randomization means that you are put into a group by chance (like flipping a coin). There is no way to predict which group you will be assigned to. You will have a one in three chance of being placed in either group. Neither you, the study staff, nor the study doctors can choose what group you will be in.

You will not know which group you are in, but the study doctor and study staff will.

WHAT IS THE STUDY INTERVENTION? Group 1: Lidocaine alone If you are randomized to this group you will receive lidocaine as your local anesthetic.

Group 2: Bupivacaine alone If you are randomized to this group you will receive bupivacaine as your local anesthetic.

Group 3: Lidocaine and bupivacaine used in combination If you are randomized to this group you will receive both lidocaine and bupivacaine used in combination during your procedure. First you will receive injections of lidocaine and then immediately afterwards you will receive injections of bupivacaine. Roughly equal volumes of lidocaine and bupivacaine will be used and the investigators expect the overall volume of local anesthetic (compared with group 1 and 2) that will be injected will be similar. The investigators expect the total number of needle pokes to be similar.

WHAT ELSE DO I NEED TO KNOW ABOUT THE STUDY INTERVENTION? All of the study interventions are considered standard of care for the use of local anesthetics in Mohs procedure. Local practices for using anesthetics are center dependent.

If you have side effects while you are on this study, the study doctor may make changes to the intervention.

If you require greater than three levels during your Mohs procedure, your data will be collected but will be excluded from the main study analysis. Patients requiring greater than three levels during their Mohs procedure are excluded because they often require more complex skin reconstruction surgery which can be more painful afterwards. The vast majority of patients undergoing Mohs surgery require one to three levels and it is these patients that the investigators are hoping to apply the results of our study to.

QUESTIONNAIRES As part of the study, you will be required to complete the same short questionnaire a total of nine times. This questionnaire will only be done by participants in this study.

The questionnaire will be completed at The Mohs Clinic just prior to your surgery and you will complete the questionnaire at home after your surgery at various time points (at 2, 4, 6, 8, 12, 24, 36 and 72 hours post surgery). The purpose of the questionnaire is assess the level of your surgical/incisional pain after Mohs surgery and enquire about any additional pain medications that you have taken after the surgery. It will take approximately 2 minutes to complete the questionnaire You will be asked to bring all of the completed questionnaires with you when you return to the Mohs Clinic for your follow-up visit one the investigatorsek after your surgery.

The information you provide is for research purposes only. You can choose not to ansthe investigatorsr questions if you wish.

Even though you may have provided information on a questionnaire, these responses will not be reviethe investigatorsd promptly by your health care team. If you wish them to know this information please bring it to their attention.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Confirmed diagnosis of non-melanoma skin cancer
3. Written informed consent

Exclusion Criteria:

1. Documented or reported history of adverse reaction to lidocaine or bupivacaine
2. Active soft tissue infection at site of surgery
3. Participants who require more than 3 stages of excision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-06-14 (Estimated)

PRIMARY OUTCOMES:
Wong-Baker FACES Pain Rating Scale | 2, 4, 6, 8, 12, 24, 36, and 72 hours
  The Wong-Baker Pain Scale is a validated tool used around the world for to quantify patients amount of pain. The score ranges from 0 (no pain) to 10 (worst pain).

SECONDARY OUTCOMES:
Adverse Event | 1 week post-op
  Adverse event to local anesthetic
Post-Operative Infection | 1 week post-op
  Post-operative infection requiring topical or systemic antibiotics
Post-Operative Bleeding | 1 week post-op
  Post-operative bleeding requiring surgical exploration/revision or hematoma evacuation

CONTACTS AND LOCATIONS:
Overall Officials: Jillian A Macdonald, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- Mohs Surgery Clinic, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bouloux GF, Punnia-Moorthy A. Bupivacaine versus lidocaine for third molar surgery: a double-blind, randomized, crossover study. J Oral Maxillofac Surg. 1999 May;57(5):510-4; discussion 515. doi: 10.1016/s0278-2391(99)90063-0. PMID 10319823
- [Result] Firoz BF, Goldberg LH, Arnon O, Mamelak AJ. An analysis of pain and analgesia after Mohs micrographic surgery. J Am Acad Dermatol. 2010 Jul;63(1):79-86. doi: 10.1016/j.jaad.2009.10.049. PMID 20542176
- [Result] Tetzlaff JE. The pharmacology of local anesthetics. Anesthesiol Clin North Am. 2000 Jun;18(2):217-33, v. doi: 10.1016/s0889-8537(05)70161-9. PMID 10935008
- [Result] Koay J, Orengo I. Application of local anesthetics in dermatologic surgery. Dermatol Surg. 2002 Feb;28(2):143-8. doi: 10.1046/j.1524-4725.2002.01126.x. PMID 11860425
- [Result] Christensen J, Matzen LH, Vaeth M, Wenzel A, Schou S. Efficiency of bupivacaine versus lidocaine and methylprednisolone versus placebo to reduce postoperative pain and swelling after surgical removal of mandibular third molars: a randomized, double-blinded, crossover clinical trial. J Oral Maxillofac Surg. 2013 Sep;71(9):1490-9. doi: 10.1016/j.joms.2013.05.001. Epub 2013 Jul 15. PMID 23866780
- [Result] Kaurich MJ, Otomo-Corgel J, Nagy RJ. Comparison of postoperative bupivacaine with lidocaine on pain and analgesic use following periodontal surgery. J West Soc Periodontol Periodontal Abstr. 1997;45(1):5-8. PMID 9477866
- [Result] Markovic AB, Todorovic L. Postoperative analgesia after lower third molar surgery: contribution of the use of long-acting local anesthetics, low-power laser, and diclofenac. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Nov;102(5):e4-8. doi: 10.1016/j.tripleo.2006.02.024. Epub 2006 Aug 10. PMID 17052624
- [Result] Su N, Liu Y, Yang X, Shi Z, Huang Y. Efficacy and safety of mepivacaine compared with lidocaine in local anaesthesia in dentistry: a meta-analysis of randomised controlled trials. Int Dent J. 2014 Apr;64(2):96-107. doi: 10.1111/idj.12087. Epub 2014 Jan 16. PMID 24428507
- [Result] Thomson CJ, Lalonde DH. Randomized double-blind comparison of duration of anesthesia among three commonly used agents in digital nerve block. Plast Reconstr Surg. 2006 Aug;118(2):429-32. doi: 10.1097/01.prs.0000227632.43606.12. PMID 16874214
- [Result] Yilmaz YF, Ozlugedik S, Titiz A, Tuncay A, Ozcan M, Unal A. Comparison of levo-bupivacaine and lidocaine for postoperative analgesia following septoplasty. Rhinology. 2008 Dec;46(4):289-91. PMID 19145998